CLINICAL TRIAL: NCT01159002
Title: Clinical Evaluation of SmartPill Capsule for Investigation of Total Intestinal Transit Time and Intestinal Pathology in Critically Ill Patients
Brief Title: Evaluation of Gastrointestinal Motility With SmartPill
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Stefan Raugh, Principal investigator, University of Louisville
Other Study IDs: SmartPill
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Gastrointestinal Motility
Keywords: Endoscopy, Video Capsule; Motility, Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically ill ICU patients: ICU patients with brain injuries who will be receiving a feeding tube.
  Interventions: Device: SmartPill

INTERVENTIONS:
Device: SmartPill — Qualifying patients were assigned to the study within four days of hospital admission. They all received a gastro-duodenal tube and capsule. The motility capsule (SmartPill®) was placed into the capsule delivery device (AdvanCE™, US Endoscopy) and advanced blindly into the stomach and released

SUMMARY:
The purpose of this study is to evaluate the clinical usefulness of a capsule (SmartPill~) measuring pH, pressure and temperature from within the entire GI tract to determine gastric emptying time, combined small and large bowel transit time and total transit time. In addition, the Capsule will characterize pressure patterns and provide motility indices for the antrum and duodenum. It is believed that the condition of your digestive system can have a large impact on your overall physical health. Therefore,the investigators would like to assess whether using the pill device helps to determine any functional problems in patients in the ICU. The investigators are studying ICU patients because any change in their condition can have a large impact on their recovery.

ELIGIBILITY:
Inclusion Criteria:

* suffered from traumatic or non-traumatic intracranial hemorrhage and were admitted to an intensive care unit (ICU) at University of Louisville Hospital
* sedated and had tracheal intubation and mechanical ventilation
* older than 18 years

Exclusion Criteria:

* younger than 18 years
* multiple injuries, especially abdominal trauma or inflammatory bowel disease
* history of complicated abdominal surgery or unknown type of abdominal surgery
* clinical evidence of ileus or suspected bowel obstruction
* a pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with intracranial hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Transit time | 5 days
  The subjects were followed from the time of placement of the capsule in the stomach until the capsule was viewed in the stool or abdominal X-rays revealed it had passed from the body

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rauch, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States